CLINICAL TRIAL: NCT04702035
Title: Walking Pattern Characteristics in Normal Pressure Hydrocephalus. A Phase I/II Open-label Single Center Trial to Characterize Disease-specific Walking Patterns Using Wearable Gyroscopes
Brief Title: Walking Pattern Characteristics in Normal Pressure Hydrocephalus
Acronym: NPH wearables
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: ETH Zurich (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NPH wearables
Record Dates: First submitted 2020-11-15; First posted 2021-01-08 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Idiopathic Normal Pressure Hydrocephalus (INPH)

STUDY DESIGN:
Intervention Model Description: Three groups of individuals are enrolled in parralel: 20 iNPH patients, 20 age- and gender-matched healthy individuals and 20 young individuals.
Masking Description: unmasked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- iNPH patients (Experimental): 20 patients with completed diagnostics concerning NPH, in which the indication for implantation of a VP shunt for NPH treatment was found by the responsible surgeon independently from the study.
  Interventions: Device: Characterization of walking pattern characteristics in an ambulatory setting using wearable IMUs (ZurichMOVE sensors)
- Healthy volunteers (Active Comparator): 20 volunteers, matched with group 1 concerning sex and age.
  Interventions: Device: Characterization of walking pattern characteristics in an ambulatory setting using wearable IMUs (ZurichMOVE sensors)
- Young healthy volunteers (Active Comparator): 20 volunteers, matched with group 1 concerning sex only and between 18 and 40 years old.
  Interventions: Device: Characterization of walking pattern characteristics in an ambulatory setting using wearable IMUs (ZurichMOVE sensors)

INTERVENTIONS:
Device: Characterization of walking pattern characteristics in an ambulatory setting using wearable IMUs (ZurichMOVE sensors) — All participants receive a set of 5 wearable IMUs for a period of 3 days. The IMUs are fixed at both wrists, ankles and one over the sternum. A 10-meter walking test, 180 degree turnaround test and normal walking at home are performed. Afterwards, the IMUs are removed for data extraction and evaluation. The patient group is examined a second time after CSF diversion surgery.

SUMMARY:
20 patients who are diagnosed with NPH receive a set of 5 wearable gyroscopes (IMUs, ZurichMove sensors) for a period of 3 days for measurement and characterization of their walking in an ambulatory setting. At a follow-up 2 weeks to 6 months after CSF diversion surgery, the examination is repeated and improvement is measured. The data will be compared with a healthy group of 20 age- and gender-matched individuals as well a a group of 20 young individuals.

DETAILED DESCRIPTION:
Temporary attachment of IMUs to wrists and ankles of the patients and probands for a period of three days and recording of movement during a 10 meter-walking test, 180° turnaround and during normal movement at home.

Group 1 (patients):

Patients with a completed diagnostic concerning iNPH, who are planned to receive a VP-shunt by their responsible neurosurgeon (independently from the study), will be included.

Before the shunt implantation, the patients will be examined at the USZ using wearable gyroscopes (like wristwatches) at both wrists and ankles as well as one around the body center.

The short examination will comprise a patient history (MoCa test, Kiefer-score, Stein- and Langfitt-Score), a short examination (4 minute walking test, 180° turnaround) in hospital. Afterwards, the patient goes home, where the gyroscopes examine walking patterns for a period of three days. After this period, the patient brings the devices back to the hospital. The surgery will take place afterwards, independently from the study, as well as adjustments of the shunt's flow-resistance for achievement of optimal response to the therapy. After this optimal result is achieved, but latest after 6 months, the examination will be repeated.

Groups 2 and 3 (controls):

As well 20 subjects matched for sex and age with the patient's group as 20 healthy young subjects will be examined just like the patients preoperatively. Walking patterns shall be compared to identify changes between pre- and postoperatively as well as differences between patients and controls.

ELIGIBILITY:
Age limits for the NPH patient group and the matched healthy vonunteers group are 60-100 years.

Age limits for the young healthy volunteers group are 18-40 years.

Inclusion Criteria:

NPH patient group:

1. Informed Consent as documented by signature prior to any study related procedures or informed consent by a legal representative in case of cognitive deficits.
2. Male and female patients alike
3. Age between 60 and 100 years
4. Clinical suspect for NPH
5. Significant improvement (by more than 10%) in walking speed or endurance in a standardized CSF-TAP test (of at least 35 ml CSF).
6. Planned implantation of a VP shunt for NPH treatment (independently from the study).

Matched controls group:

1. Informed Consent as documented by signature prior to any study related procedures
2. Male and female patients alike (matched to group 1)
3. Age between 60 and 100 years (matched to group 1)
4. No clinical suspect for NPH or any other movement disorder

Young controls group:

1. Informed Consent as documented by signature prior to any study related procedures
2. Male and female patients alike (matched to group 1)
3. Age between 18 and 40 years
4. No clinical suspect for NPH or any other movement disorder

Exclusion Criteria:

1. Enrolment of the investigator, his/her family members, employees and other dependent persons (only for patients; no exclusion criteria for controls),
2. Apparent or suspected movement disorder or other known disorder, which might affect normal standing or walking
3. Cardiovascular disorders, which might affect physical resilience
4. Pregnant women
5. Pre-menopausal state of female patients and probands in groups 1 and 2.
6. Children and adolescents

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2024-04-25 (Actual); Study Completion 2024-04-25 (Actual)

PRIMARY OUTCOMES:
Walking characteristics | Between 2 weeks to 6 months after CSF diversion surgery
  Complex walking pattern comprising of stride length, width, frequency (altogether one parameter)

SECONDARY OUTCOMES:
4 minutes timed Walk test | immediately after fixation of IMUs
  Standard test (seconds)
180 degree turnaround test | immediately after fixation of IMUs
  Participants are asked to turn by 180 degrees. Steps needed are counted.
Kiefer score | before surgery
  Standard score for iNPH severity, only patient group; range 0-26; higher indicates higher severity
Kiefer score | after surgery (range 2 weeks to 6 months)
  Standard score for iNPH severity, only patient group; range 0-26; higher indicates higher severity
Stein and Langfitt score | before surgery
  Standard score for patient independence, only patient group; range 0-IV; higher indicates higher dependency
Stein and Langfitt score | after surgery (range 2 weeks to 6 months)
  Standard score for patient independence, only patient group; range 0-IV; higher indicates higher dependency
NPH recovery rate | after surgery (range 2 weeks to 6 months)
  Standard rate for success of CSF diversion treatment in NPH. Calculated as follows: (Kiefer score preoperatively - Kiefer score postoperatively) / Kiefer score preoperatively x 10; range 0-10; Higher indicates better response to surgery
Evan´s Index | before surgery
  Standard descriptor for width of lateral ventricles in iNPH. Calculated as maximum with of frontal horns / maximal diameter of brain in axial CT or MRI at the level of cella media; range: 0-1; higher indicates larger ventricles and more severe hydrocephlaus
Disproportionally Enlarged Subarachnoidal space Hydrocephalus (DESH) sign | before surgery
  Positivity of standard sign in preoperative CT or MRI imaging, hinting at presence of iNPH. Values: Positive/Negative
Time from appearance of first symptoms to surgery | before surgery
  From first appearance of symptoms to surgery in years
3-dimensional characterization of walking patterns | before surgery
  Detailed analysis of walking patterns recorded during the measurement phases by the wearable IMUs.
3-dimensional characterization of walking patterns | after surgery (range 2 weeks to 6 months)
  Detailed analysis of walking patterns recorded during the measurement phases by the wearable IMUs.

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of Neurosurgery, Zurich University Hospital, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No
Sharing of data with other researchers is not intended.

REFERENCES:
- [Background] Renggli D, Graf C, Tachatos N, Singh N, Meboldt M, Taylor WR, Stieglitz L, Schmid Daners M. Wearable Inertial Measurement Units for Assessing Gait in Real-World Environments. Front Physiol. 2020 Feb 20;11:90. doi: 10.3389/fphys.2020.00090. eCollection 2020. PMID 32153420